CLINICAL TRIAL: NCT07072975
Title: CPOD Patient's Tolerance of Intermittent Exercise With Inter-exercise Recovery Under Normoxic Hypoxia
Acronym: HypoChronoPerf
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2025_843_0029
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Intermittent Hypoxia; Exercise Recovery; Intermittent Exercise; Rating Exertion Perception; Sleep
Keywords: intermittent hypoxia; exercise recovery; intermittent exercise; rating exertion perception; sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- comparator (Experimental): On separate days, 50 patients with COPD completed four sets of 4-min at 85% of VO2peak intercept by 3-min of passive recovery in two randomized between-sets recovery conditions. Rating exertion perception, gaz exchanges, heart rate, sleep quality and nocturnal heart rate variability were assessed.
  Interventions: Other: Normobaric hypoxia
- sham (Sham Comparator)
  Interventions: Other: normoxic condition

INTERVENTIONS:
Other: Normobaric hypoxia — Normobaric hypoxia (inspired oxygen fraction of 12.9%) applied between-sets recovery periods
  Arms: comparator
Other: normoxic condition — Between-sets recovery periods under normoxic condition
  Arms: sham

SUMMARY:
Exercise retraining improves the prognosis and quality of life of patients with chronic lung or circulatory diseases. However, exercise intolerance may be caused by excessive ventilatory. Exposure to oxygen-replete air reduces this ventilatory overload, improves sleep and enhances responses to exercise. This study examine the impact of the acute manipulation of oxygen availability during inter-exercise recovery period of an intermittent cycling exercise on perceptual responses.

this randomized, controlled, study include adult patient with COPD. On separate days, 50 patients with COPD completed four sets of 4-min at 85% of VO2peak intercept by 3-min of passive recovery in two randomized between-sets recovery conditions. Rating exertion perception, gaz exchanges, heart rate, sleep quality and nocturnal heart rate variability were assessed.

Hypoxic exposure during inter-repetition recovery phases would reduce the ventilatory load during exercise. What's more, patients would not be forced to perform the sporting gesture in a restricted space or wearing a mask, limiting dyspnea and the perceived difficulty of the effort. Lastly, the induction of hypoxic stress during the re-training session helped to improve patients' sleep.

ELIGIBILITY:
Inclusion Criteria:

* from 40 to 60 years
* follow-up in the pneumology unit of CHU Amiens - Picardie
* Chronic Obstructive Pulmonary Disease stade II
* Body mass index from 20 to 30 kg.m-2
* Tiffeneau index < 70% of predicted value
* FEV1 from 50 to 80% of predicted values
* Smoking cessation since at least 1 week
* Sedentary or physical active
* Affiliate to social security
* Written consent

Exclusion Criteria:

-

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Perception Exertion score with CR10 | day 1
  The modified Borg CR10 RPE scale measures exertion on a scale of 0 (no exertion or resting) to 10 (pushing yourself to the max).

SECONDARY OUTCOMES:
Cardiorespiratory responses to exercise | day 1
  Cardiorespiratory responses to exercise is measured with gaseous exchange volumes

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No